CLINICAL TRIAL: NCT07305571
Title: The Effect of Psychodrama-Based Group Work on Postpartum Women's Depression and Forgiveness Tendencies: A Randomised Controlled Study
Brief Title: The Effect of Psychodrama-Based Group Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ömer USLU (Other)
Responsible Party: Sponsor-Investigator, Ömer USLU, Dr. Ömer Uslu, PhD - Principal Investigator, Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MERVE-RCT-2025-PAD
Record Dates: First submitted 2025-12-13; First posted 2025-12-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Psychiatric Nursing; Depression Disorder; Forgiveness; Puerperal Depression; Psychoeducation
Keywords: depression; forgiveness; psychodrama; puerperal; psychiatric nursing
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Intervention Model Description: This study used a pretest-posttest-follow-up randomised controlled experimental method. Participants were randomly assigned to either the experimental group (psychodrama-based group intervention) or the control group with no intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- psychodrama-based group intervention (Experimental): Participants will receive an 8-session psychodrama-based group intervention.
  Interventions: Other: psychodrama-based group intervention; Other: Control
- Control (No Intervention): Throughout the study, the psychodrama-based group intervention was applied only to the experimental group, and no intervention was performed in the control group

INTERVENTIONS:
Other: psychodrama-based group intervention — For postpartum mothers in the experimental group, a psychodrama-based group intervention was carried out face-to-face, with one session per week, each lasting 120 minutes, for a total of 8 sessions (over 8 weeks).
  Arms: psychodrama-based group intervention
Other: Control — no intervention was performed in the control group
  Arms: psychodrama-based group intervention

SUMMARY:
Aims This study examined the effect of psychodrama-based group work on postpartum women's tendencies toward depression and forgiveness.

Methods This study used a pretest-posttest-follow-up randomised controlled experimental method. The study sample consisted of 23 postpartum mothers (11 experimental and 12 control) whose babies were receiving treatment in the neonatal intensive care unit between April and June 2025. While psychodrama-based group intervention was applied to the experimental group, no intervention was performed in the control group. Data were collected using a personal information form, Postnatal Depression Screening Scale, and Forgiveness Scale.

Results In the study, it was found that the mean forgiveness scores in the final test and follow-up measurements of the postpartum women in the experimental group were statistically significantly higher compared to the control group (p<0.05). In the final test and follow-up measurements, the mean postpartum depression scores of the women in the experimental group were found to be statistically significantly lower than those of the mothers in the control group (p<0.05).

Conclusions Psychodrama-based group work increased forgiveness tendencies and reduced depression levels in postpartum women. In this regard, it is recommended that psychodrama sessions be conducted for postpartum women.

DETAILED DESCRIPTION:
The neonatal period is a critical stage of development in the first 28 days after birth, during which the baby adapts physiologically and biologically to the external environment. Owing to issues such as prematurity, low birth weight, congenital anomalies, and respiratory distress, some babies require advanced medical support, highlighting the vital importance of the Neonatal Intensive Care Unit (NICU). During this process, mothers experience intense psychological stress due to factors such as uncertainty about the baby's health, limited physical contact, a highly technological environment, and the postponement of maternal roles, which leads to the emergence of negative emotions, such as guilt, inadequacy, hopelessness, helplessness, and anxiety, thereby making the postpartum period more emotionally fragile. These negative emotions also weaken the psychological resilience of postpartum mothers and constitute a significant risk factor, especially for the development of postpartum depression. Studies in the literature indicate that mothers experiencing postpartum depression negatively affect their breastfeeding behaviors, adaptation to the postpartum period, ability to cope with challenges, quality of life, and overall mental, physical, and social health. The concept of forgiveness, which facilitates relief from pain and distress caused by intense negative emotions that intensify during the postpartum period, is defined as an important psychological component in overcoming depression, anxiety, relationship conflicts, and crises in a healthy manner. Forgiveness has been reported to make a significant contribution, particularly in reducing depressive symptoms. Forgiveness has been shown to have positive effects in alleviating psychological distress, protecting and improving health, and has been found to be beneficial in the treatment of various mental disorders. One such approach is psychodrama. Psychodrama has been used in the field of nursing since the 1960s and has found a place in clinical practice. Psychodrama is an effective and important psychotherapy method in terms of increasing peer support, finding a model for identification, experiencing positive relationships, seeing different approaches to relationships, and experiencing different roles. An increase in the number of psychiatric nurses with knowledge and skills in psychodrama will add a scientific and artistic dimension to the field of nursing, creating a special level of advancement in the quality of care provided by nurses through interactions with people. In this context, considering the critical role of women in shaping the future of society, this study evaluated the effects of a psychodrama-based group intervention aimed at supporting the psychological well-being of mothers during the postpartum period, reducing depressive symptoms, and strengthening tendencies toward forgiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-55 years or (until menopause)
* Having the mental capacity and sufficient communication skills to follow the research instructions, being literate.
* Having an infant receiving treatment in the neonatal intensive care unit.

Exclusion Criteria:

* Having a condition that impairs communication
* Having a diagnosed mental illness.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-06-29 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Postpartum Depression Screening Scale | Baseline (pretest), 8 weeks (posttest) and one month after the posttest
  Evaluation of the change in the total score of the Postpartum Depression Screening Scale. The minimum score obtained from the scale was 35, and the maximum score was 175. Higher scores indicate higher levels of postpartum depression.

SECONDARY OUTCOMES:
The Forgiveness Scale | Baseline (pretest), 8 weeks (posttest) and one month after the posttest
  Forgiveness Scale, developed by Ersanlı and Batık, designed to measure individuals' levels of self-forgiveness and forgiveness of others. The scale is scored from "strongly disagree" to "strongly agree," with higher scores indicating higher levels of forgiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Şahin, PhD, RN, Principal Investigator — Bergama Necla Mithat Öztüre State Hospital
Locations (1):
- Bergama Necla Mithat Öztüre State Hospital, Izmir, Bergama, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared due to ethical and institutional restrictions. The dataset includes sensitive health information from postpartum women, and the informed consent process did not include permission for public data sharing. Therefore, in accordance with privacy regulations and ethical committee requirements, IPD will not be made available to other researchers

REFERENCES:
- See also: Bergama Necla Mithat Öztüre State Hospital — https://bergamadh.saglik.gov.tr